CLINICAL TRIAL: NCT06633536
Title: Real-life Treatment Outcomes of Ravulizumab in Polish Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH). Prospective and Retrospective, Multicenter, Non-interventional Study.
Brief Title: Real-life Treatment Outcomes of Ravulizumab in PNH
Acronym: PNH-RECORD
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9289R00001
Record Dates: First submitted 2024-08-09; First posted 2024-10-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Haemoglobinuria
Keywords: Paroxysmal nocturnal haemoglobinuria; PNH; ravulizumab
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ravulizumab group: Open-label
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — open-label arm with ravulizumab administrated within the scope of routine clinical practice

SUMMARY:
The PNH-RECORD study, a Polish multicenter observational (non-interventional), open-label, retrospective with prospective follow-up.

DETAILED DESCRIPTION:
PNH-RECORD study aims to aims to collect data on the patients' characteristics and clinical outcomes of ravulizumab administered in the scope of routine clinical practice in PNH.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged ≥18) patients with PNH receiving ravulizumab treatment in the frames of NDP in Poland.
2. Patients willing to participate in the study and signed ICF.

Exclusion Criteria:

1. Those who participated in ravulizumab clinical trial in the past, and/or those who participated/plans to participate in clinical trial on/after the date of first ravulizumab infusion through NDP.
2. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (aged ≥18) patients with PNH
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in LDH levels from index date (first dose of ravulizumab) at every 6 month | up to 36 months
Proportion of patients achieving or remaining at LDH<1.5 ULN at every 6 month | up to 36 months

SECONDARY OUTCOMES:
Proportion of transfusion-free patients from index date at every 6 month | up to 36 months
Number of blood units used per patient-year | up to 36 months
To present patients characteristics | Baseline
  Mean age (years) at PNH diagnosis
To present patients characteristics | Baseline
  Mean age (years) at index date
To present patients characteristics | Baseline
  Proportion (%) of men and women
To present patients characteristics | Baseline
  Mean body mass index (kg/m²)
To present clinical characteristics | Baseline
  Mean and median (years) duration of PNH
To present clinical characteristics | Baseline
  Mean and median (months) time from diagnosis to complement inhibitors treatment initiation
To present clinical characteristics | Baseline
  Proportion (%) of patients with complication of haemolysis, thrombosis, serious vascular event andaplastic anemia
To present clinical characteristics | Baseline
  Proportion (%) of patients naïve to complement inhibitors

CONTACTS AND LOCATIONS:
Locations (11):
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Brzozów
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wałbrzych

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/